CLINICAL TRIAL: NCT04932928
Title: Patient-Driven Lifestyle Modification Using FreeStyle Libre in Type 2 Diabetes Patients
Acronym: PDF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Inje University (Other); Kangbuk Samsung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2011-062-117
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Lifestyle Risk Reduction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FreeStyle Libre (CGM) Group (Experimental): Device: FreeStyle Libre (ver 1.0) Education on lifestyle modification
  Interventions: Device: FreeStyle Libre
- Self Monitoring of Blood Glucose (SMBG) Group (Active Comparator): Device: Blood glucose meter Education on lifestyle modification
  Interventions: Device: Blood glucose meter

INTERVENTIONS:
Device: FreeStyle Libre — Flash glucose monitoring + Education on lifestyle modification
  Other Names: Education on lifestyle modification
  Arms: FreeStyle Libre (CGM) Group
Device: Blood glucose meter — Self monitoring of blood glucose + Education on lifestyle modification
  Other Names: Education on lifestyle modification
  Arms: Self Monitoring of Blood Glucose (SMBG) Group

SUMMARY:
We aim to provide medical nutritional therapy to patients with type 2 diabetes who are on oral hypoglycemic agents or on basal insulin only and monitor the glycemic response with flash glucose monitoring or self-monitoring of blood glucose.

Specifically, this is a randomized, open-label, controlled study where half of the study participants will have FreeStyle Libre device on for 12 weeks and compare the change in glycated hemoglobin (HbA1c) value with the patients in the control group.

DETAILED DESCRIPTION:
Subjects: 126 patients with type 2 diabetes mellitus Scheme: Multi-center, Randomized, open-label, controlled study

This study is referred to as the "Patient-Driven lifestyle modification using FreeStyle Libre in type 2 diabetes patients", also known as the PDF study.

It will assess potential benefits of using Continuous Glucose Monitoring (CGM) versus Self Monitoring of Blood Glucose (SMBG) when combined with personalized education on lifestyle modification in people with type 2 diabetes. Specifically, we will investigate patients who have an elevated HbA1c between 7.0 - 10.0% who are not using prandial insulin.

Potential participants will be screened from routine outpatient clinic visits, will be randomized to either the CGM or SMBG group in a 1:1 ratio. Participants from both groups will receive education on lifestyle modification and will be reminded every 4 weeks with structured phone visits. Study will be completed at the visit on 12 weeks of follow up with the same laboratory examinations (including HbA1c) and survey from the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80
* Diagnosed with type 2 diabetes mellitus (DM)
* Uncontrolled type 2 DM: HbA1c 7.0-10.0%
* Signed informed consent

Exclusion Criteria:

* Diagnosed with other types of diabetes mellitus (i.e. Type 1 DM)
* Use of prandial insulin
* Change in diabetes medication in the preceding 3 months
* Pregnant/lactating women
* Addiction to drugs and alcohol
* Use of medications that result in drug-induced hyperglycemia (i.e. steroid)
* Severe liver disease
* End-stage renal disease (i.e. on dialysis)
* Unable to wear CGM devices due to dermatologic side effects (i.e. severe burn, inflammation, active skin infection, severe skin reactions, hypertrichosis, etc.)
* Conditions that impact the stability of HbA1c measurement

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-09-23 (Estimated); Study Completion 2023-03-23 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in HbA1c from baseline to Month 3

SECONDARY OUTCOMES:
Change in mean fasting glucose | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in fasting glucose from baseline to Month 3
Change in body weight | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in body weight from baseline to Month 3
Change in blood pressure | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in blood pressure from baseline to Month 3
Change in waist circumference | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in waist circumference from baseline to Month 3
Change in lipid level | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in lipid level (total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol) from baseline to Month 3
Change in the Korean Version of Revised Summary of Diabetes Self-Care Activities Questionnaire (SDSCA-K) survey score | Baseline to Month 3
  Between group differences (CGM and SMBG) for the change in survey score from baseline to Month 3

OTHER OUTCOMES:
Change in CGM time in target range | Baseline to Month 3
  Change in CGM time in target range 70-180 mg/dL from baseline to Month 3 in the CGM group
Change in CGM time-hyperglycemic | Baseline to Month 3
  Change in CGM time in time above target range, defined as >250 mg/dL from baseline to Month 3 in the CGM group
Change in CGM time-hypoglycemic | Baseline to Month 3
  Change in CGM time in time below target range, defined as <70 mg/dL (level 1) and < 54 (level 2) from baseline to Month 3 in the CGM group
Change in CGM glucose variability | Baseline to Month 3
  Change in CGM glucose variability measured by the coefficient of variation from baseline to Month 3 in the CGM group

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choe HJ, Rhee EJ, Won JC, Park KS, Lee WY, Cho YM. Effects of Patient-Driven Lifestyle Modification Using Intermittently Scanned Continuous Glucose Monitoring in Patients With Type 2 Diabetes: Results From the Randomized Open-label PDF Study. Diabetes Care. 2022 Oct 1;45(10):2224-2230. doi: 10.2337/dc22-0764. PMID 35984640